CLINICAL TRIAL: NCT06335368
Title: Assessment of Nutritional and Growth Status in Rett Syndrome Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201512178RINC
Record Dates: First submitted 2022-07-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2022-07

CONDITIONS: Rett Syndrome; Neurologic Disorder
MeSH Terms: conditions — Rett Syndrome; Nervous System Diseases | interventions — Nutritional Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nutrition and Growth Status — Nutrition and Growth Status

SUMMARY:
Children with Rett syndrome are in a period of rapid growth, and proper and appropriate nutritional support is very important. Past foreign research papers it has been pointed out that most of these patients have feeding difficulties, dysphagia, and digestive tract abnormalities, are often constipated, and may suffer from osteoporosis and other problems. Lack of proper nutritional support will seriously affect their growth, development and health. in view of There is a lack of relevant research in China, so the investigators would like to use this research to explore the nutritional, growth and postural status of Rett's disease patients, as the reference direction and goal of dietary adjustment and nutritional support for patients, and establish dietary and nutritional strategies for sick children in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Rett syndrome patient.

Exclusion Criteria:

* Not Rett syndrome patient.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Rett syndrome patient.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2016-05-23 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
gender, age , disease history checklist | 1 year
Change in Body height | 1 year
  The growth status of the case will be assessed
Change in Body weight | 1 year
  The growth status of the case will be assessed
Change in knee height | 1 year
  The growth status of the case will be assessed
Change in arms height | 1 year
  The growth status of the case will be assessed and growth curve
Change in waist | 1 year
  The growth status of the case will be assessed
Change in hip circumferences | 1 year
  The growth status of the case will be assessed

IPD SHARING:
Plan to Share IPD: No
Assessment of nutritional and growth status in Rett syndrome patient